CLINICAL TRIAL: NCT04641533
Title: Effect of Dental Pulp Stem Cells and L-PRF Placed Into the Extraction Sockets of Impacted Mandibular Third Molars on the Periodontal Status of Adjacent Second Molars: a Split Mouth Randomised Controlled Clinical Trial
Brief Title: Effect of Dental Pulp Stem Cells and L-PRF After Impacted Third Molar Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Secil Cubuk, Assist Prof, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SecilC
Record Dates: First submitted 2020-08-16; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Stem Cell; Third Molar; Periodontal Pocket
Keywords: dental pulp; stem cell; third molar; Platelet-rich fibrin
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Intervention Model Description: Prospective within person randomised split-mouth study. Left and right surgical sites for each participant were randomized using an online generated list to determine test and positive control LM3. (http://www.randomization.com). LM2s and LM3 extraction sockets were divided into two groups: a test group (extraction sockets filled with L-PRF membranes + DPSCs) and a control group (extraction sockets filled with L-PRF membranes).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The random allocation list was generated by a periodontist (EEA), a clinical staff enrolled patients according to their reference date. The first allocation on the list was assigned to the right mandibular molar for each patient by the oral surgeon (SÇ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF + DPSC (Experimental): Mandibular third molars were extracted and DPSC with L-PRF placed into the socket.
  Interventions: Procedure: L-PRF + DPSC
- L-PRF (Active Comparator): Mandibular third molars were extracted and L-PRF placed into the socket
  Interventions: Procedure: L-PRF

INTERVENTIONS:
Procedure: L-PRF + DPSC — After surgical removal of impacted mandibular third molars, extraction sockets were filled with L-PRF membranes + DPSCs.
  Other Names: Leukocyte platelet rich fibrin plus dental pulp stem cells
  Arms: L-PRF + DPSC
Procedure: L-PRF — After surgical removal of impacted contralateral mandibular third molars, each extraction sockets were only filled with L-PRF membranes.
  Other Names: Leukocyte platelet rich fibrin
  Arms: L-PRF

SUMMARY:
The purpose of this study is to compare the clinical and radiographic effectiveness of Leukocyte-Platelet Rich Fibrin (L-PRF) and L-PRF combined with dental pulp stem cell (DPSC) application to the extraction socket of mandibular third molars.

DETAILED DESCRIPTION:
Patients aged between 18 and 30 years, seeking for bilateral impacted LM3 extraction surgeries and meeting eligibility criteria were included to the study. At baseline right and left impacted third molars (LM3s) were randomly assigned to one of the treatment group (L-PRF and L-PRF + DPSC). Baseline and 6th month clinical and radiographic measurements were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 30 years
* Bilateral impacted LM3 extraction surgeries requirement

Exclusion Criteria:

* Having clinical signs or symptoms of abscess or cellulitis formation
* Having a history of radiotherapy
* Having any systemic diseases interfering with wound healing and/or smokers
* Patients who had been diagnosed as periodontitis
* Patients who had LM2s with caries or restorations that have an unidentifiable cementoenamel junction

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Probing pocket Depth (PPD) | 6 months
  Probing pocket Depth (PPD) is the distance between gingival margin and bottom of the periodontal pocket in mm.
Clinical attachment level (CAL) | 6 months
  Clinical attachment level (CAL) is the distance between cemento-enamel junction and bottom of the periodontal pocket in mm.

SECONDARY OUTCOMES:
Radiographic vertical distance | 6 months
  The cementoenamel junction (CEJ) and the most coronal point of the alveolar bone were identified (AC) on the mesial and distal of lower second molars on digital panoramic radiographs. The vertical ruler on each digital image was used to calibrate the image and to convert measurements from pixels to millimeters with ImageJ. The vertical distance (VD) between cemento-enamel junction and alveolar crest of the lower second molar was than measured with "straight line" tool of the software. In order to calculate the real distance; ertical distance was divided to the magnification factor for panoramic image (1.2).
Relative bone density (rBD) | 6 months
  For every extraction socket, a region of interest (ROI) is created for the socket region and one for the surrounding bone using the "Freehand Selection" tool of ImageJ software on panoramic radiographs. Mean grey values were recorded for each group and relative bone density (rBD) was calculated.
Post-operative pain as assessed by visual analogue scale (VAS) | 7 days
  Self-reported pain measured in a 100 mm visual analogue scale (VAS) in which (0) denoted "no pain" and 100 meant "severe pain" was recorded at the end of the surgery and 7 days after extraction.
Assessment of analgesic usage | 7 days
  The patients were asked to note the amount of analgesics within the post-operative 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Alaaddinoğlu, Prof,PhD, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cubuk S, Oduncuoglu BF, Alaaddinoglu EE. The effect of dental pulp stem cells and L-PRF when placed into the extraction sockets of impacted mandibular third molars on the periodontal status of adjacent second molars: a split-mouth, randomized, controlled clinical trial. Oral Maxillofac Surg. 2023 Mar;27(1):59-68. doi: 10.1007/s10006-022-01045-2. Epub 2022 Feb 9. PMID 35141806